CLINICAL TRIAL: NCT04966039
Title: Diffusion Weighted Magnetic Resonance Imaging of Brain in Monochorionic Twin Pregnancies With Demise of One Fetus
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017316
Record Dates: First submitted 2021-06-29; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Twin Pregnancy With Antenatal Problem
Keywords: twin pregnancy; demise of one fetus; Diffusion weighted imaging; Diffusion tensor imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- monochorionic twin pregnancies with demise of one fetus: Twin pregnancy was diagnosed and one fetus died in utero, 20 pregnant women
  Interventions: Other: No intervention.
- Twin control group: Twin pregnancy with one abnormal fetus, 20 pregnant women
  Interventions: Other: No intervention.
- Singleton control group: Singleton pregnancy with abnormalities outside the fetal brain, 20 pregnant women
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — There was no intervention.

SUMMARY:
Diffusion weighted imaging (DWI) can reflect the microstructure and pathological changes of tissue, and diffusion tensor imaging (DTI) can quantitatively evaluate the fine structure of white matter in brain. In this study, conventional and diffusion-weighted MRI (DWI, DTI) sequences were used to analyze the brain of monochorionic twin pregnancies with demise of one fetus.

DETAILED DESCRIPTION:
With the incidence rate of twin pregnancy increasing, the incidence of intrauterine death of twin pregnancies is also rising, which has great impact on the morbidity and mortality of the other fetus, and increases the mortality of fetal survival, premature birth, brain damage and long-term sequela. Therefore, it is necessary to examine the central nervous system of the surviving fetus of twin pregnancy and intrauterine death. When the surviving fetus is complicated with nervous system abnormalities, conventional MRI can generally make a diagnosis. However, some of the surviving fetuses may not find other structural or echo abnormalities on B-mode ultrasonography, and even these fetuses do not find structural or signal abnormalities on routine MRI examination. Whether the surviving fetuses may have brain abnormalities cannot be detected early by the above methods. Diffusion weighted imaging (DWI) can reflect the microstructure and pathological changes of tissue, and diffusion tensor imaging (DTI) can quantitatively evaluate the fine structure of white matter in brain.

The present study is to use conventional sequence and diffusion-weighted imaging (DWI, DTI) to analyze the brain of monochorionic twin pregnancies with demise of one fetus, which aims to find the potential brain abnormalities early and provide some guidance for the clinical diagnosis and treatment in the next step.

ELIGIBILITY:
Inclusion Criteria:

1. Twin pregnancy was diagnosed and one fetus died in utero
2. Twin pregnancy with one abnormal fetus
3. Singleton pregnancy with abnormalities outside the fetal brain

Exclusion Criteria:

1. Those who can't cooperate with MRI examination, such as those who have metal, claustrophobia or can't insist on scanning.
2. Pregnant women with gestational age less than 20 weeks.

Age Groups: Child, Adult, Older Adult
Study Population: 1. Twin pregnancy was diagnosed and one fetus died in utero
  2. Twin pregnancy with one abnormal fetus
  3. Singleton pregnancy with abnormalities outside the fetal brain
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
basic information | baseline
  age
basic information | baseline
  gestational age
basic information | baseline
  uterine height
basic information | baseline
  abdominal circumference
basic information | baseline
  intrauterine death time of one fetus
MRI | baseline
  DWI sequence (ADC value)
MRI | baseline
  DTI sequence (FA value)
MRI | baseline
  conventional sequence

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China